CLINICAL TRIAL: NCT04717362
Title: The Effects of Natesto For Treatment Of Hypogonadism On Maintenance Of Spermatogensis.
Brief Title: The Effects of Natesto For Treatment Of Hypogonadism
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No longer wanting to enroll or start study.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Larry I. Lipshultz, rofessor of Urology and Chief of the Scott Department of Urology's Division of Male Reproductive Medicine and Surgery, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48763
Record Dates: First submitted 2020-12-07; First posted 2021-01-22 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Hypogonadism, Male; Infertility, Male; Testosterone Deficiency
Keywords: Natesto; Male; Hypogonadism; Sexual Medicine
MeSH Terms: conditions — Eunuchism; Infertility, Male; Hypogonadism

STUDY DESIGN:
Intervention Model Description: Prospective non-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard Reboot with Natesto (Experimental): Standard Reboot Protocol + Natesto
  Interventions: Drug: Natesto Nasal Product

INTERVENTIONS:
Drug: Natesto Nasal Product — Nasally administered exogenous 4.5% testosterone gel, administered from a non-pressurized, manual pump dispenser equipped with a specialized nasal applicator which administers 125uL (5.5mg of testosterone).

SUMMARY:
In this prospective study, the investigators plan is to confirm the role of Natesto (intranasal testosterone) to combat hypogonadal symptoms in men trying to recover spermatogenesis following the withdrawal of conventional Testosterone replacement therapy.

DETAILED DESCRIPTION:
Testosterone replacement therapy (TTh) is becoming increasingly common among men of reproductive age in the United States. An estimated 3 million men are on TTh; however exogenous testosterone use can disrupt the hypothalamus-pituitary-gonadal (HPG) axis, leading to reduced spermatogenesis and possible infertility. In normal physiology, the hypothalamus releases Gonadotropin-releasing hormone (GnRH), which stimulates the anterior pituitary to release Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH). FSH then stimulates the Sertoli cells in the testis to support spermatogonial differentiation and maturation. LH stimulates the Leydig cells in the testes to produce endogenous testosterone. Regulation of this HPG axis occurs via negative feedback where testosterone directly inhibits the release of GnRH and LH from the hypothalamus and pituitary, respectively. The use of exogenous testosterone thus leads to reduced Sertoli function causing diminished spermatogenesis.

The spontaneous recovery of spermatogenesis after cessation of TTh is possible but may take months to years and cause the patient to experience new onset of severe hypothalamic hypogonadal symptoms. Human chorionic gonadotropin (HCG) is a naturally occurring protein that mimics LH and may be used as a therapy to support the return of spermatogenesis quickly with minimal side effects and resolve hypogonadal symptoms. Studies have shown that testosterone-induced infertile patients can recover sperm in the ejaculate in 4.6 months when treated with HCG supplemented with clomiphene citrate, tamoxifen, anastrozole, or recombinant FSH. With the cessation of TTh, despite the use of LH stimulatory protocols, these patients still experience hypogonadal symptoms. Recent preliminary results show the potential to offset hypogonadism symptoms that accompany exogenous testosterone cessation through administration of 4.5% intranasal testosterone gel. Natesto is a nasally administered exogenous 4.5% testosterone gel, administered from a non-pressurized, manual pump dispenser equipped with a specialized nasal applicator which administers 125uL (5.5mg of testosterone). Previous studies have shown that a single nasal dose has a rapid absorption with a Tmax at 60 mins and a half-life that ranged between 10-100 minutes. Three to four daily doses achieve eugonadal levels of circulating testosterone comparable to normal pulsatile-regulated release of testosterone. It has also been shown that men on Natesto maintain FSH and LH levels as well as total motile sperm count within the normal range. In this prospective study, the investigators seek to confirm the role of Natesto to combat hypogonadal symptoms in men trying to recover spermatogenesis following the withdrawal of conventional TTh.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily sign and date the study consent form(s) which have been approved by an Institutional Review Board (IRB). Written consent must be obtained prior to the initiation of any study procedures.

  2. Male between 18 and 64 years of age, inclusive, with documented onset of testosterone induced hypogonadism with impaired semen parameters who are attempting to achieve a successful pregnancy.

  3. Documented diagnosis of primary hypogonadism (congenital or acquired) or hypogonadotropic hypogonadism (congenital or acquired).

  4. Serum total testosterone < 350 ng/dL based on 2 consecutive blood samples obtained 1-4 weeks apart between 6 and 10 AM following an appropriate washout of current androgen replacement therapy; with clinical symptoms of hypogonadism such as diminished energy and sexual function; and/or a decreased sperm count (<20 million sperm/mL semen).

  5. Discontinued current testosterone replacement treatment and completed a washout of 4 weeks following androgen treatment (excluding Testopel TM). Washout must be completed prior to collection of baseline serum testosterone samples to determine study eligibility.

  6. Judged to be in good general health as determined by the principal investigator based upon the results of a medical history, physical examination, vital signs, and laboratory profile.

Exclusion Criteria:

* 1. History of significant sensitivity or allergy to androgens, castor oil or product excipients.

  2. Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up.

  3. Abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or I-PSS score > 19 points.

  4. Body mass index (BMI) ≥ 35 kg/m2.

  5. History of vasectomy.

  6. Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:
  1. Baseline hemoglobin > 16 g/dL
  2. Hematocrit < 35% or > 50%
  3. PSA > 4 ng/mL and age >40

     7. History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.

     8. History of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study drug administration.

     9. History of stroke or myocardial infarction within the past 5 years.

     10. History of, or current or suspected, prostate or breast cancer.

     11. History of diagnosed, severe, untreated, obstructive sleep apnea.

     12. History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.

     13. History of nasal disorders such as nasal polyps; nasal septal perforation; nasal surgery; nasal trauma resulting in nasal fracture within the previous 6 months or nasal fracture that caused a deviated anterior nasal septum; sinus surgery or sinus disease

     14. Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 12 weeks prior to the start of treatment.

     15. Inadequate venous access for collection of serial blood samples required for pharmacokinetic profiles.

     16. Receipt of any investigational product within 4 weeks or within 5 half-lives prior to the start of treatment.

     17. Inability to understand and provide written informed consent for the study.

     18. Considered by the investigator or the sponsor-designated physician, for any reason, that the subject is an unsuitable candidate to receive Natesto.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Semen Analysis | Baseline, 14 weeks, 26 weeks.
  Change in Total Motile Sperm

SECONDARY OUTCOMES:
Change in Hypogonadal Panel | Baseline, 14 weeks, 26 weeks.
  change in blood LH levels
Change in Hypogonadal Panel | Baseline, 14 weeks, 26 weeks.
  change in blood FSH levels
Change Hypogonadal Panel | Baseline, 14 weeks, 26 weeks.
  change in blood Testosterone levels
Change in Hypogonadal Panel | Baseline, 14 weeks, 26 weeks.
  change in blood E2 levels
Change in Quality of Life Questionnaire | Baseline, 14 weeks, 26 weeks.
  Change in SF36 score
Change in Quality of Life Questionnaire | Baseline, 14 weeks, 26 weeks.
  Change in IPSS score
Change in Quality of Life Questionnaire | Baseline, 14 weeks, 26 weeks.
  Change in IIEF score

IPD SHARING:
Plan to Share IPD: No